CLINICAL TRIAL: NCT04420663
Title: Pleural Manometry During Thoracocentesis in Patients With Malignant Pleural Effusion: How Much Fluid Should we Drain?
Brief Title: Pleural Manometry in Thoracocentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aly Sherif Hassaballa (Other)
Responsible Party: Sponsor-Investigator, Aly Sherif Hassaballa, Clinical Professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ASHassaballaMD
Record Dates: First submitted 2020-04-15; First posted 2020-06-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Thoracocentesis of Pleural Effusion

STUDY DESIGN:
Intervention Model Description: This prospective controlled trial study will be performed between August 2019 and August 2020. We will enroll patients with large volume pleural effusion referred to our Cardiothoracic Department, Faculty of Medicine, Ain Shams University to perform therapeutic thoracentesis. All the patients will sign an informed consent for pleural pressure monitoring during and after therapeutic thoracentesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manometer Group (Experimental): Therapeutic thoracentesis will be performed in a sitting position. wide bore catheter as a pleural catheter will be inserted into the pleural cavity. simple water manometer will be connected to the pleural catheter via 3-way adapter.connected to the infusion lines with one draining into the drainage collection bottle and the other pre-flushed with normal saline hanging down till 40 cm below the puncture site and then rising up (forming a "U") with the ascending arm taped to the IV stand. baseline pleural pressure will be registered before the beginning of pleural fluid withdrawal. Pleural pressure curve will subsequently be registered after the withdrawal of each 200 ml of pleural fluid up to a total volume of 1000 ml.
  Interventions: Diagnostic Test: Pleural Manometry
- Conventional Group (No Intervention): Therapeutic thoracentesis will be performed in a sitting position. The skin will be cleaned with betadine antiseptic solution. Pleural aspiration should take place in a clean area using full aseptic techniques. 5-10 cc Lidocaine 2% will be given as local anesthetic in the site of puncture. the IV cannula is advanced till fluid is aspirated. Then, the needle is withdrawn and the catheter is fixed to two 3-way adapters fixed in series placed in between. connected to the infusion lines with one draining into the drainage collection bottle.

INTERVENTIONS:
Diagnostic Test: Pleural Manometry — Recording pleural pressure during therapeutic thoracocentesis using a simple water manometer.
  Arms: Manometer Group

SUMMARY:
The study aiming to measure the pleural pressure during thoracocentesis in patients with pleural effusion and the value of their measurement in both diagnostic and therapeutic decisions.

DETAILED DESCRIPTION:
This prospective controlled trial study will be performed between July 2019 and December 2020. the investigators will enroll patients with large volume pleural effusion referred to our Cardiothoracic Department, Faculty of Medicine, Ain Shams University to perform therapeutic thoracentesis. All the patients will sign an informed consent for pleural pressure monitoring during and after therapeutic thoracentesis.

The study aiming to measure the pleural pressure during thoracocentesis in patients with pleural effusion and the value of their measurement in both diagnostic and therapeutic decisions.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 85 years,
2. pleural effusion occupying at least one-third of the ipsilateral hemithorax in P-A chest radiograph (CXR)
3. no contraindications for therapeutic thoracentesis
4. general health condition allowing prolonged procedure of therapeutic thoracentesis.

Exclusion Criteria:

* patients with very small amounts of pleural effusion
* patients on mechanical ventilation
* patients using anticoagulant therapy
* patients refusing to be subjected to thoracocentesis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
the pleural pressure | Continous monitoring during the whole session of thoracocentesis
  To measure the pleural pressure(mmHg) during thoracocentesis in patients with pleural effusion using a simple water pleural manometer

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiothoracic Surgery Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassaballa AS, Mostafa A, Hikal T, Elnori A, Elsayed HH. Pleural manometry during thoracocentesis in patients with malignant pleural effusion: A randomized controlled trial. Can J Respir Ther. 2023 Jan 20;59:33-44. doi: 10.29390/cjrt-2022-047. eCollection 2023. PMID 36741303